CLINICAL TRIAL: NCT06467422
Title: Exploring the Role and Neural Mechanisms of Transcranial Temporal Interference Stimulation Modulating the Dorsal Anterior Cingulate Cortex on Risky Decision-making and Impulse Control in Gambling Disorder
Brief Title: Effects of Transcranial Temporal Interference Stimulation on Risky Decision-making and Impulse Control in Gambling Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MZhao-017
Record Dates: First submitted 2024-06-06; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theta Stimulation(6Hz, generated with electrodes of 2kHz and 2.005kHz) (Experimental): Session1#T1(10min)+DTI(15min) Session2#rsfMRI(8min)+rsfMRI-Theta tTIs(8min)+rsfMRI(8min)+TASK fMRI-Theta TI(20min)
  Interventions: Device: tTIS on dACC, theta frequency (5 Hz)
- High Frequency Stimulation(generated with two electrodes of 2kHz) (Sham Comparator): Session1#T1(10min)+DTI(15min) Session2#rsfMRI(8min)+rsfMRI-HF tTIs(8min)+rsfMRI(8min)+TASK fMRI-HF TI(20min)
  Interventions: Device: tTIS on dACC, High frequency

INTERVENTIONS:
Device: tTIS on dACC, theta frequency (5 Hz) — Device: Transcranial electric stimulation device
  The first pair of electrodes continuously outputs a current with a frequency of f1 = 2 kHz, while the second pair continuously outputs a current with a frequency of f2 = 2.006 kHz. According to the principle of time-domain coherence, an alternating electric field with a frequency of f2-f1 = 6 Hz can be generated in the target area. The experimental group receives a stimulation intensity of 2mA for 20 minutes. The optimal electrode position and current parameters are determined by using the MIDA head electric field model.
  Arms: Theta Stimulation(6Hz, generated with electrodes of 2kHz and 2.005kHz)
Device: tTIS on dACC, High frequency — The first pair of electrodes continuously outputs a current with a frequency of f1 = 2 kHz, while the second pair continuously outputs a current with a frequency of f2 = 2 kHz. The sham group receives a stimulation intensity of 2mA for 20 minutes. The optimal electrode position and current parameters are determined by using the MIDA head electric field model.
  Arms: High Frequency Stimulation(generated with two electrodes of 2kHz)

SUMMARY:
The purpose of this research is to investigate the effect of transcranial temporal interference stimulation (tTIS) targeting the dorsal anterior cingulate cortex in patients with gambling disorder.

DETAILED DESCRIPTION:
This study will apply the emerging non-invasive deep brain stimulation of tTIS to the dorsal anterior cingulate cortex in a randomized, double-blind design to demonstrate the possibility of non-invasively targeting the anterior cingulate cortex to modulate impulse control and risky decision-making without activating other regions below the electrodes. Additionally, this study will combine the fMRI recordings to describe local and network effects on brain activity. Specifically, each participant will be assessed at baseline with a scale and T1WI sequence and diffusion tensor imaging, and will randomly receive a combination of stimulation sequentially during the intervention phase, with more than a one-week interval ensuring that there is no interference between each of the two stimulation sequences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60, male or female, right handed;
* With 9 or more years of education, and able to cooperate in completing the questionnaire assessment and behavioural tests.
* Meets the DSM-5 diagnostic criteria for gambling addiction;
* Previous gambling behaviour of not less than 1 year's duration (at least one gambling session per week or more);
* Normal or corrected normal vision and hearing;
* Agrees to cooperate in completing the follow-up assessment;
* No history of neurological problems or head injury; and no skin sensitivity.
* Agree to cooperate in completing the follow-up assessment;
* No metal implantation in the head, no history of neurological problems or head injury, and no skin sensitivity.

Exclusion Criteria:

* Suffering from severe cognitive dysfunction, such as a history of head trauma, cerebrovascular disease, epilepsy, etc., use of cognitive-promoting medications in the last 6 months;
* Other psychoactive substance abuse or dependence in the last 5 years (except nicotine).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Activation of dACC | Through the fMRI procedure
  Activation of dACC is measured with resting-state fMRI and task fMRI.
Activation of decision-making network | Through the fMRI procedure
  Activation of decision-making network is measured with resting-state fMRI and task fMRI connectivity analysis.
The change of impulsivity | Through the last 20 minutes of the fMRI session.
  The change of impulsivity will be measured by sequential decision-making task.

SECONDARY OUTCOMES:
The change of gambling craving | 8 minutes, 16 minutes, 24 minutes, 44 minutes of the fMRI session.
  Gambling craving will be measured by the gambling craving Visual Analog Scale (VAS). The total score of VAS ranged from 0 to 10, in which higher scores mean a higher level of gambling craving.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, M.D, Ph.D, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided